CLINICAL TRIAL: NCT01540201
Title: The Effect of Different I:E Ratio on Gas Exchange of Patients Undergoing One-lung Ventilation for Lung Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Sangmin M. Lee, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2011-12-033-002
Record Dates: First submitted 2012-02-16; First posted 2012-02-28 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Lung Cancer; One Lung Ventilation; Gas Exchange; Inverse-ratio Ventilation
Keywords: one lung ventilation; gas exchange; inverse-ratio ventilation
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1:2 group (Active Comparator): conventional I:E ratio group, inspiratory time : expiratory time = 1:1
  Interventions: Other: Conventional I:E ratio
- 1:1 group (Experimental): inspiratory time : expiratory time = 1:1
  Interventions: Other: I:E = 1:1 ratio

INTERVENTIONS:
Other: Conventional I:E ratio — conventional I:E ratio of 1:2 is applied. Ventilator : Datex-Ohmeda Aestiva/5 ® model
  Other Names: I:E ratio of 1:2; Ventilator : Datex-Ohmeda Aestiva/5 ® model
  Arms: 1:2 group
Other: I:E = 1:1 ratio — I:E ratio of 1:1 is applied Ventilator : Datex-Ohmeda Aestiva/5 ® model
  Other Names: I:E ratio of 1:1; Ventilator : Datex-Ohmeda Aestiva/5 ® model
  Arms: 1:1 group

SUMMARY:
Pulmonary gas exchange disturbance is a common anesthetic problem during one-lung ventilation (OLV) for thoracic surgery. The inverse-ratio ventilation (IRV), which prolongs the inspiratory time greater than expiratory time, can be applied for adult respiratory distress syndrome. The effect of IRV is to improve gas-exchange status by increasing mean airway pressure and alveolar recruitment. We tried to evaluate the effect of IRV during OLV with lung protective strategy.

DETAILED DESCRIPTION:
Pulmonary gas exchange disturbance is a common anesthetic problem during one-lung ventilation (OLV) for thoracic surgery. Continuous positive airway pressure or positive end-expiratory pressure are usually applied to improve this disorder including hypoxia, but these methods are not enough. The inverse-ratio ventilation (IRV), which prolongs the inspiratory time greater than expiratory time, can be applied for adult respiratory distress syndrome. The effect of IRV is to improve gas-exchange status by increasing mean airway pressure and alveolar recruitment. The application of IRV during OLV has not been performed to our knowledge, and there is a possibility of IRV to improve oxygenation during OLV. There is a possibility of increase of auto-PEEP, or air trapping in subjects with chronic obstructive pulmonary disease, but this kind of auto-PEEP can be overcome by external PEEP. Therefore, we tried to evaluate the effect of IRV during OLV with lung protective strategy.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective lung lobectomy surgery.
* the duration of one-lung ventilation is more than one hour.
* subjects with more than twenty years old.

Exclusion Criteria:

* subjects with past history of pneumothorax, asthma
* Age under 20, more than 70 years.
* Patients with ischemic heart disease, valvular heart disease
* patients with hemodynamic unstability

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
arterial CO2 partial pressure | 10 minutes after induction of general anesthesia
  arteial CO2 partial pressure
arterial CO2 partial pressure | 30 minutes after start of one-lung ventilation
  arteial CO2 partial pressure
arterial CO2 partial pressure | 60 minutes after start of one-lung ventilation
  arteial CO2 partial pressure
arterial CO2 partial pressure | 15 min after restart of TLV
  arteial CO2 partial pressure
arterial CO2 partial pressure | 1 hour after the end of surgery
  arteial CO2 partial pressure

SECONDARY OUTCOMES:
arterial O2 partial pressure | 10 min after induction, 30 and 60 min after start of one-lung ventilation, 15 min after restart of two-lung ventilation, 1 hour after the end of surgery
  arterial O2 partial pressure
Mean airway pressure | 10 min after induction, 30 and 60 min after start of one-lung ventilation, 15 min after restart of two-lung ventilation
  Mean airway pressure
tidal volume (exhaled) | 10 min after induction, 30 and 60 min after start of one-lung ventilation, 15 min after restart of two-lung ventilation
  tidal volume (exhaled)
hemodynamic parameters | 10 min after induction, 30 and 60 min after start of one-lung ventilation, 15 min after restart of two-lung ventilation
  systolic/ diastolic blood pressure, heart rate, mean blood pressure
end-tidal CO2 partial pressure | 10 min after induction, 30 and 60 min after start of one-lung ventilation, 15 min after restart of two-lung ventilation
  end-tidal CO2 partial pressure
respiratory compliance | 10 min after induction, 30 and 60 min after start of one-lung ventilation, 15 min after restart of two-lung ventilation
  Dynamic compliance, Static compliance
Dead space | 10 min after induction, 30 and 60 min after start of one lung ventilation, 15 min after restart of two-lung ventilation
  physiologic dead space / tidal volume (VD/VT)
work of breathing | 10 min after induction, 30 and 60 min after start of one-lung ventilation, 15 min after restart of two-lung ventilation
  work of breathing
peak inspiratory pressure | 10 min after induction, 30 and 60 min after start of one-lung ventilation, 15 min after restart of two-lung ventilation
  peak inspiratory pressure
plateau pressure | 10 min after induction, 30 and 60 min after start of one-lung ventilation, 15 min after restart of two-lung ventilation
  plateau pressure
positive end-expiratory pressure | 10 min after induction, 30 and 60 min after start of one-lung ventilation, 15 min after restart of two-lung ventilation
  positive end-expiratory pressure
minute ventilation | 10 min after induction, 30 and 60 min after start of one-lung ventilation, 15 min after restart of two-lung ventilation
  minute ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Sangmin M. Lee, MD, PhD, Principal Investigator — Samsung Medical Center; Won Ho Kim, MD, Study Director — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea